CLINICAL TRIAL: NCT04463992
Title: Lay Health Worker Expanded Intervention in Community Oncology Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 57643
Record Dates: First submitted 2020-07-04; First posted 2020-07-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: End of Life; Cancer
Keywords: cancer end of life patient-centered
MeSH Terms: conditions — Death; Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group Arm (Experimental): Patients randomized into the intervention will be assigned a lay health worker who will contact the patient to begin the intervention. The intervention includes: proactive symptom assessments for patients for up to 12-months.
  Interventions: Behavioral: Program participants; Other: Usual Care
- Behavioral:Program participants (Active Comparator): The control group arm will receive usual care as provided by their local oncologists.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Program participants — The intervention is a 12-month telephonic program in which a lay health worker (LHW), supervised on-site by a registered nurse practitioner (RNP), assessed patient symptoms after diagnosis using the validated Edmonton Symptom The intervention is a 12-month telephonic program in which a lay health worker (LHW), supervised on-site by a registered nurse practitioner (RNP), assessed patient symptoms after diagnosis using the validated Edmonton Symptom Assessment Scale (ESAS) (cite) with the frequency of symptom assessment varying based on patient risk.
  Arms: Intervention Group Arm
Other: Usual Care — Usual care as provided by local oncologists

SUMMARY:
Undertreated patient symptoms and resulting acute care use require approaches that improve symptom-burden. Previously a lay health worker (LHW)-led symptom screening intervention was developed for patients with cancer. In pilot work, the intervention was associated with improvements in patient symptom burden and reductions in healthcare use and costs of care at the end of life. This intervention will be expanded across several clinics to evaluate the impact of the LHW intervention on with cancer and the LHW will be trained to refer patients to palliative care. This randomized intervention will evaluate the effect on healthcare use, total costs, palliative care and hospice referral.

DETAILED DESCRIPTION:
All patients with newly diagnosed cancer, over the age of 75 will be randomized into the CareMore Pilot 2 Program with 200 randomized to the intervention grou and 200 randomized to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or relapsed cancer diagnosis.
* 75 years or older
* Diagnosis of relapse or progressive disease (any cancer diagnosis) as identified by imaging or biopsy and confirmed by physician.
* Must have capacity to verbally consent

Exclusion Criteria:

* Inability to consent to the study due to lack of capacity as documented by the referring physician.

Ages: 75 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 416 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
% of patients with Emergency Department Visit within 12-months after patient enrollment (Chart Review) | 12 months after patient enrollment
  Emergency Department use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment. We will evaluate comparisons of the % of patients with emergency department visits between study arms.
% of patients with Hospitalization Visits within 12 months after patient enrollment (Chart Review) | 12 months after patient enrollment
  Hospitalization use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment. We will evaluate comparisons of hospitalizations between the two study arms.

SECONDARY OUTCOMES:
% of patients with a Hospice Consult within 12-months after patient enrollment (Chart Review) | 12 months after patient enrollment
  Hospice consult for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.
Total Health Care Costs (Claims Review) | 12 months after patient enrollment
  Total Health Care Costs for each patient will be abstracted by medical claims data review for each patient at 12 months after enrollment.
% of patients with an Acute Care Facility Death (Chart Review) | 30 days prior to death for patients who died at 12-months follow-up
  Acute Care Facility Deaths for each patient will be abstracted by electronic medical record chart review and claims review for each patient who has died at 12-months followup. We will evaluate comparisons of Acute Care Facility Deaths between study arms.
% of patients with Emergency Department Visit in the last 30 days of life (Chart Review) | 30 days prior to death for patients who died at 12-months follow-up
  Emergency Department use for each patient will be abstracted by electronic medical record chart review for each patient who has died. We will evaluate comparisons of emergency department visits between study arms.
% of patients with Hospitalization Visits in the last 30 days of life (Chart Review) | 30 days prior to death for patients who died at 12-months follow-up
  Hospital use for each patient will be abstracted by electronic medical record chart review for each patient who has died. We will evaluate comparisons of hospitalization use between study arms.
% of patients with a Hospice Consult in the last 30 days of life (Chart Review) | 30 days prior to death for patients who died at 12-months follow-up
  Hospice use for each patient will be abstracted by electronic medical record chart review for each patient who has died. We will evaluate comparisons of hospice use between study arms.
Total Costs of Care (Claims Review) | Time of enrollment to 12 months followup or death, whichever is first
  Total costs of care for each patient will be obtained through claims data for each patient for each patient who has died. We will evaluate comparisons of Total costs of care between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Manali I Patel, MD MPH MS, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - The Oncology Institute of Hope and Innovation, Tucson, Arizona
  - The Oncology Institute of Hope and Innovation, Henderson, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel MI, Voskanyan M, Agajanian H, Agajanian R, Podnos Y, Milstein A. A Lay Health Worker-Led Symptom Intervention and Acute Care Use in Older Adults With Cancer: A Randomized Clinical Trial. JAMA. 2025 Dec 30:e2523403. doi: 10.1001/jama.2025.23403. Online ahead of print. PMID 41468027